CLINICAL TRIAL: NCT06415669
Title: A Study of Paclitaxel (Albumin-bound) Combined With Apatinib and Adebrelimab in the Treatment of Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma Following Previous Immunotherapy Progression
Brief Title: A Study of Paclitaxel Combined With Apatinib and Adebrelimab in Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Mingquan Cai, Director of medical oncology, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-FJ-GC-II-013
Record Dates: First submitted 2024-04-27; First posted 2024-05-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma
Keywords: paclitaxel; apatinib; adebrelimab; adenocarcinoma of the gastroesophageal junction; gastric carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Injections; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Paclitaxel for injection (albumin-bound) in combination with Apatinib mesylate and adebrelimab
  Interventions: Drug: Paclitaxel for injection (albumin-bound); Drug: Adebrelimab; Drug: Apatinib mesylate

INTERVENTIONS:
Drug: Paclitaxel for injection (albumin-bound) — 100 mg/m2, day 1, day 8, every 21 days for a cycle.
Drug: Adebrelimab — 20mg/kg or 1200mg, the first day, every 21 days as a cycle.
  Other Names: SHR-1316
Drug: Apatinib mesylate — 250mg once a day for 5 consecutive days and discontinue for 2 days

SUMMARY:
To evaluate the initial efficacy and safety of paclitaxel for injection (albumin-bound) in combination with apatinib mesylate and adebrelimab in the treatment of locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma following the progression of previous immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18 ~ 75 years old, male and female;
* 2) ECOG score: 0 or 1;
* 3) Patients with unresectable locally advanced or metastatic gastric cancer/gastroesophageal junction adenocarcinoma confirmed by histopathology;
* 4) Patients who have received at least first-line immunotherapy progression or intolerance in the past, and the number of previous systemic treatment lines does not exceed 2 lines; The best curative effect of frontline containing PD-1/PD-L1 was CR, PR or SD;
* 5) According to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1), there should be at least one measurable lesion that has not received local treatment such as radiotherapy (lesions located in the area of previous radiotherapy can also be selected as target lesions if progression is confirmed);
* 6) The major organs function normally and meet the following criteria
* a. In the past 14 days without the use of granulocyte colony-stimulating factor, the absolute value of neutrophil (ANC) ≥1.5x109 /L;
* b. Platelets ≥100×109 /L in the past 14 days without blood transfusion;
* c. Hemoglobin >90g/L in the last 14 days without blood transfusion or use of erythropoietin;
* d. Total bilirubin ≤1.5× upper limit of normal (ULN);
* e. aspartate aminotransferase (AST), alanine aminotransferase (ALT) in

  ≤2.5×ULN (ALT or AST ≤5×ULN for patients with liver metastasis);
* f. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥40 ml/min;
* g. Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
* h. The myocardial enzyme profile is within the normal range (if the researchers comprehensively judge that the simple laboratory abnormality is not clinically significant, it is also allowed to be included);
* 7) Expected survival ≥3 months;
* 8) Women of reproductive age should agree to use contraceptives (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient; Men should consent to patients who must use contraception during the study period and for 6 months after the end of the study period;
* 9) Sign informed consent.

Exclusion Criteria:

* 1) Patients who have previously received paclitaxel chemotherapy; Patients with neoadjuvant or adjuvant treatment with taxoid drugs and disease progression more than 6 months after the last chemotherapy were excluded;
* 2) HER2-positive patients;
* 3) Patients who are taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone) and continue to use within 2 weeks before enrollment;
* 4) Patients with severe liver and kidney insufficiency or heart insufficiency;
* 5) have multiple factors that affect oral drugs (such as inability to swallow, gastrointestinal resection, chronic diarrhea, and intestinal obstruction);
* 6) Patients with brain metastases accompanied by symptoms or symptom control for less than 3 months;
* 7) Patients who are known to be allergic to any investigational drug or drug excipient;
* 8) Pregnant or lactating female patients;
* 9) Patients who underwent major surgical procedures (craniotomy, thoracotomy, or laparotomy) or had unhealed surgical wounds, ulcers, or fractures within 4 weeks prior to initial dosing, except for patients ≥2 weeks after surgery and patients with old fractures that the investigator determined could be treated with the study drug;
* 10) Patients with moderate to severe ascites accompanied by clinical symptoms requiring repeated drainage; Patients with uncontrolled or clinical symptoms of pleural effusion or pericardial effusion;
* 11) Patients with clinically significant electrolyte disorders;
* 12) People with acute or chronic active hepatitis B or hepatitis C: hepatitis B virus (HBV) DNA > 2000IU/ml or 104 copies /ml; Hepatitis C virus (HCV) RNA > 103 copies /ml; Hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive patients;
* 13) Patients with central nervous system metastasis, but with no clinical symptoms or accompanied by clinical symptoms after treatment, disease control and stable time ≥4 weeks can be enrolled; To meet the need for measurable lesions outside the central nervous system, hormone therapy should be discontinued 14 days before the first study of medication
* 14) Any life-threatening bleeding event within the previous 3 months, including patients requiring transfusion therapy, surgery or local therapy, and ongoing medication;
* 15) Patients with a history of arteriovenous thromboembolism events, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other severe thromboembolism within the past 6 months. The exception is implantable intravenous infusion port or catheter-derived thrombosis, or superficial venous thrombosis, which is stable after conventional anticoagulant therapy. Allow patients to prophylactically use small doses of low molecular weight heparin (e.g., enoxaparin 40 mg/ day);
* 16) Uncontrolled hypertension, systolic blood pressure > 160 MMHG or diastolic blood pressure > 100mmHg after optimal medical treatment, hypertensive crisis or hypertensive encephalopathy history;
* 17) Symptomatic congestive heart failure (New York Heart Association Grade II-IV). Symptomatic or poorly controlled arrhythmia. Patients with a history of congenital long QT syndrome or a QTc > 500ms (calculated using the Fridericia method) corrected at screening;
* 18) For patients who received radiation therapy more than 4 weeks before the first treatment, all of the following conditions must be met to be enrolled: there is no current toxic reaction related to radiation therapy, no need to take glucocorticoids, and radiation pneumonia, radiation hepatitis, and radiation enteritis are excluded;
* 19) Patients with previous or current pulmonary diseases such as pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severe impairment of lung function;
* 20) Human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive), known syphilis infection;
* 21) Patients with unhealed wounds, fractures, gastric and duodenal ulcers, persistent positive stool occultiblood, ulcerative colitis, or other conditions that researchers have determined may cause gastrointestinal bleeding or perforation;
* 22) All adverse events during the screening period have not returned to baseline or ≤ Grade 1 (NCI-CTCAE V5.0) (except for alopecia, or peripheral sensory neuropathy, which can be grade 2);
* 23) Patients with severe infections that are active or poorly controlled clinically. Patients with severe infections in the 4 weeks prior to initial dosing, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia;
* 24) Use of immunosuppressive drugs within 4 weeks prior to initial administration, excluding nasal, inhaled, or other routes of topical corticosteroids or physiological doses of systemic corticosteroids (i.e., no more than 10mg/ day of prednisone or equivalent doses of other corticosteroids); To allow temporary use of glucocorticoids for the treatment of breathing difficulties in diseases such as asthma and chronic obstructive pulmonary disease;
* 25) Patients who received live attenuated vaccine within 4 weeks prior to initial administration or who planned to receive live attenuated vaccine during the study period;
* 26) Patients who received major surgical treatment or significant traumatic injury 4 weeks prior to initial dosing
* 27) Patients who received traditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first dose;
* 28) Patients with a history of gastrointestinal perforation or abscess within 6 months prior to enrollment;
* 29) Received treatment in other clinical trials within 4 weeks prior to initial dosing;
* 30) Patients whose urine routine indicated urinary protein ≥2+, or 24-hour urinary protein quantity >1.0g;
* 31) The presence of any active autoimmune disease or history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis); Patients with asthma requiring medical intervention with bronchodilators were not included); However, the following patients were admitted: vitiligo, psoriasis, alopecia, well-controlled type I diabetes without systemic therapy, hypothyroidism with normal thyroid function treated by replacement therapy;
* 32) Other acute or chronic medical conditions, psychiatric disorders, or abnormalities in laboratory test values that may contribute to these results: increase the risk associated with study participation or study drug administration, or interfere with the interpretation of study results, and, in the investigator's judgment, classify patients as ineligible to participate in the study;
* 33) Other situations deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 1 years
  Refers to the proportion of all subjects with the best overall response (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Disease control rate（DCR） | 1 years
  Refers to the proportion of all subjects with the best overall response (BOR) according to RECIST1.1 criteria as complete remission (CR), partial remission (PR) and stable disease (SD).
Progression-free survival (PFS) | 1 years
  PFS was defined as the subject's date from the date of the first dose to the date of the first documented tumor progression (as assessed by RECIST1.1 criteria, with or without continuation of treatment) or the date of death from any cause, whichever occurred first.
Duration of response (DoR) Duration of response (DoR) Duration of response (DoR) Duration of response (DoR) Duration of response (DoR) Duration of response (DoR) | 1 years
  It refers to the time between the first evaluation of a tumor as CR or PR and the second evaluation as Progressive Disease (PD) or death from any cause.
Overall survival（OS） | 2 years
  Defined as the time from the date of the first dose to the death of the subject from any cause.
Occurence of AE and SAE | 2 years
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Appraisal of life quality | 1 years
  Quality of life scale for cancer patients(The EORTC's QLQ-C30 (V3.0)) is a core scale for all cancer patients with 30 entries.Items 29 and 30 are divided into seven grades, ranging from 1 to 7 according to their answer choices; Other items are rated on a four-point scale,with a straightforward scale of 1 to 4.Except for items 29 and 30, they are all reverse entries (the larger the value, the worse the quality of life).The score for each field is obtained by adding and dividing the scores for the items included in each field by the number of items included (RS).The standard component of the computing function area also changes direction. Specifically, it is calculated according to the following formula (where R is the score range of each field or item).Functional area: SS=[1-(RS-1)/R]*100 Symptom domain and general health status domain :SS=[(RS-1)/R]*100

OTHER OUTCOMES:
Explore potential biomarkers in tumor tissue | 1 years
  ORR corresponding to PD-L1 negative expression, positive expression (TPS≥1%), low expression (<10%), high expression (TPS>50%)

CONTACTS AND LOCATIONS:
Overall Officials: Mingquan Cai, Principal Investigator — The First Affiliated Hospital of Xiamen University; Xia Lv, Principal Investigator — Xiamen Humanity Hospital; Jun Qiu, Principal Investigator — Xiamen Humanity Hospital; Huita Wu, Principal Investigator — Zhongshan Hospital Affiliated to Xiamen University; Xiuping Zhang, Principal Investigator — Zhongshan Hospital (Xiamen), Fudan University; Xiaojian Yin, Principal Investigator — Xiamen Changgeng Hospital; Jinfeng Zhu, Principal Investigator — Quanzhou First Hospital; Wen Chen, Principal Investigator — The Second Affiliated Hospital of Fujian Medical University; Yijun Wang, Principal Investigator — Zhangzhou Hospital; Guoqin Qiu, Principal Investigator — The 73rd Army Hospital; Yongmei Liu, Principal Investigator — West China Xiamen Hospital of Sichuan University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No